CLINICAL TRIAL: NCT05622383
Title: Music Concert and Inhaler Aromatherapy Applied to Patients Who Have Had Coronary Angiography
Brief Title: The Effect of Music Concert and Inhaler Aromatherapy Applied to Patients Who Have Had Coronary Angiography on Pain Severity, Anxiety and Fear Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, gülcan bahcecioğlu, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022/ 10- 35
Record Dates: First submitted 2022-11-11; First posted 2022-11-18 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Anxiety; Pain
Keywords: coronary angiography; aromatherapy; music concert
MeSH Terms: conditions — Anxiety Disorders; Pain | interventions — Aromatherapy

STUDY DESIGN:
Intervention Model Description: aromatherapy, music concert
Who Masked: Participant
Masking Description: aromatherapy, music concert
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- aromatherapy (Experimental): aromatherapy will be applied
  Interventions: Other: aromatherapy
- music concert (Experimental): music concert will be applied
  Interventions: Other: music concert
- aromatherapy,music concert (Experimental): aromatherapy, music concert will be applied
  Interventions: Other: aromatherapy and music concert,
- control (No Intervention): Routine maintenance will be applied.

INTERVENTIONS:
Other: aromatherapy — aromatherapy,
  Arms: aromatherapy
Other: music concert — music concert
  Arms: music concert
Other: aromatherapy and music concert, — aromatherapy and music concert,
  Arms: aromatherapy,music concert

SUMMARY:
Coronary angiography; It is defined as the imaging of the coronary arteries by providing the catheterization of the femoral, brachial or radial arteries, and the administration of contrast material under the guidance of fluoroscopy. Coronary angiography is a stressful procedure for the patient. Because patients are conscious during the procedure, they may experience anxiety about possible complications and an uncertain outcome. Anxiety causes changes in the physiological parameters of individuals by affecting the sympathetic nervous system of individuals. As with all procedures performed in the hospital environment, patients may experience pain during coronary angiography. Coronary angiography causes fear of death and anxiety in patients due to the unknowns it contains. Aromatherapy is the use of oils obtained from plants for treatment and care. Aromatherapy provides control of pain and anxiety by affecting the amygdala and hippocampus, which regulate fear and aggression behaviors in the limbic system. Music has been used by different civilizations throughout history for purposes such as reinforcing religious feelings, intensifying emotions and curing diseases. The multifaceted effect of music on people has led to its use in treatment. Among the therapeutic benefits of listening to music are the reduction of fear, pain and anxiety by diverting the attention of the individual, affecting the autonomic nervous system and increasing the secretion of endorphins. The aim of this study is to examine the effects of aromatherapy and music listening on pain, anxiety and fear in patients who will undergo coronary angiography

DETAILED DESCRIPTION:
This study, which was planned as an experimental study with a pretest-posttest control group, will be a study for patients who will undergo coronary angiography in the angiography unit of Fırat University Hospital and Fethi Sekin City Hospital. Prior to the study, a priori power analysis was performed to determine the sample size in this study. In the power analysis, it was determined that a total of at least 120 samples, including 1st Group 30, 2nd Group 30, 3rd Group 30 and control group 30, should be at 0.05 significance level, 95% confidence interval, 95% power and 5% margin of error. Random numbers table will be used to determine the experimental and control groups. Then, by drawing lots, 1.2.3. experimental group and control group will be assigned. The patients in the experimental group will be divided into three as those who will be treated only with music, who will be treated with aromatherapy only through inhalation, and those who will be treated with music and inhalation aromatherapy together. Before any intervention is made in the intervention group and control group, the Patient Information Form, Visual Analog Scale-Pain (VAS-P), Visual Analog Scale-Fear (VAS-F), Visual Analog Scale was given to the patients to determine the pain, anxiety and fear level of these patients. -Anxiety (VAS-A), State-Trait Anxiety Inventory (DSÖ) will be used to pre-test. Inhaler aromatherapy, music concert, music concert and inhaler aromatherapy applications will be applied to the patients in the intervention groups before and during the procedure, while the control group will not receive any intervention. With the post-test, VAS-P, VAS-F, VAS-A, DSÖ will be applied to both the intervention and control groups and their pain, anxiety and fear levels will be evaluated. Finally, it will be checked whether there is a significant difference between the pre-test and post-test.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old

  * Ability to communicate adequately
  * Absence of psychiatric problems
  * Absence of an obstacle to smell
  * Volunteering to participate in the research
  * No sedation before and during the procedure
  * No known allergy to the essential oils to be applied.
  * Volunteering to participate in the research

Exclusion Criteria:

Those who have communication problems

* Those with psychiatric problems
* Having a history of allergies
* Having a known allergy to the essential oils to be applied
* Having a condition that prevents smelling
* Being uncomfortable with the smell to be applied

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2023-02-25 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale-Pain | 1 hours later
  Visual Analog Scale is used to convert some values that cannot be measured numerically into digital. Two end definitions of the parameter to be evaluated are written at the two ends of a 100 mm line and the patient is asked to indicate where on this line their situation is appropriate by drawing a line or by placing a dot or pointing.0 points means no pain, 100 points means a lot of pain
Visual Analog Scale - fear | 1 hours later
  Patients are asked to show the intensity of fear on a 10 cm long vertical or horizontal line during activity or rest. It has numbered shapes ranging from 1-10. The line has 0 at the beginning and 10 at the end. 10 means unbearable fear, 0 means no fear. The VAS scale is frequently used in the evaluation of fear severity. While the patient marks the fear he/she has felt on this line, each point he/she has marked is measured in cm.
Visual Analog Scale - Anxiety | 1 hours later
  Patients are asked to show the intensity of anxiety on a 10 cm long horizontal line during activity or rest. The line has 0 at the beginning and 10 at the end. 10 means unbearable pain, 0 means no pain. VAS is frequently used in the evaluation of pain intensity. While the patient marks the anxiety he has felt on this line, each point he has marked is measured in cm.
State-Trait Anxiety Scale | 1 hours later
  In this study, the part of the scale measuring trait anxiety was used to determine the trait anxiety levels of the patients. Trait Anxiety Inventory is a 4-point Likert-type with 20 items and is scored as "never": 1, "a little": 2, "a lot": 3, "completely": 4, according to the degree of severity of the feelings, thoughts or behaviors expressed by the items. . There are direct or reverse scored statements in the scale. Reverse scored statements; Items 1, 6, 7, 10, 13, 16 and 19. Trait anxiety score is obtained by adding the constant value of 35, which is the constant value of the trait anxiety scale, to the value obtained by subtracting the total score of the reverse scored statements from the total score of the direct statements. The lowest score that can be obtained from the scale is 20, and the highest score is 80. A high score indicates a high level of anxiety, a low score indicates a low level of anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Gülcan B Turan, Elâzığ, Merkez, Turkey (Türkiye)